CLINICAL TRIAL: NCT03340220
Title: Phase 1, First-in-human, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and PK of Single and Multiple Ascending Oral Doses of XEN1101 and Preliminary Open-label Pharmacodynamic Assessment in Healthy Subjects Addendum: Phase 1, Randomised, Multi Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Relative Bioavailability and Food Effect of Single and Multiple Ascending Doses of XEN1101 and Preliminary Drug-Drug Interaction Assessment With Itraconazole
Brief Title: Safety, Tolerability, and Pharmacokinetics (PK) of Single and Multiple Ascending Oral Doses of XEN1101.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XPF-008-101a; 2017-003168-11 (EudraCT Number); C17030 (Other: Richmond Pharmacology Ltd)
Record Dates: First submitted 2017-10-31; First posted 2017-11-13 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — microcrystalline cellulose; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Drug: XEN1101 XPF-008 Formulation Oral (Experimental): XEN1101 XPF-008 Formulation Part 1 - Single ascending dose: Single oral dose for each cohort Part 2 - Multiple ascending dose: 7 days of single oral dose daily for each cohort
  Interventions: Drug: XPF-008
- Placebo - Microcrystalline cellulose oral (Placebo Comparator): Part 1- Single Ascending Dose: Single oral dose for each cohort
  Part 2 - Multiple Ascending Dose: 7 days of single oral dose daily for each cohort
  Interventions: Drug: Microcrystalline Cellulose
- Drug: XEN1101 XPF-008 Formulation Oral Drug: XEN1101 XPF-010 Formulation Oral (Experimental): XEN1101 XPF-008 and XPF-010 Formulation Cross Over
  Part 3 will explore dose proportionality of XPF-010 and confirm dosing for subsequent cohorts, and the food effect and relative bioavailability of XPF-010 compared to XPF-008
  Interventions: Drug: XPF-010
- Drug: XEN1101 XPF-010 Formulation Oral (Experimental): XEN1101 XPF-010 Formulation Oral
  Part 4 will explore multiple dose PK
  Interventions: Drug: XPF-010
- Drug: XEN1101 XPF-010 Formulation Oral Drug: Itraconazole 400mg Oral (Experimental): XEN1101 XPF-010 Formulation + Itraconazole
  Part 5 will explore the drug-drug interaction of XPF-010, when given with itraconazole (400mg, single dose, oral solution, fasted)
  Interventions: Drug: Itraconazole 400mg

INTERVENTIONS:
Drug: XPF-008 — Capsule filled with XEN1101
  Arms: Drug: XEN1101 XPF-008 Formulation Oral
Drug: Microcrystalline Cellulose — Placebo capsule
  Arms: Placebo - Microcrystalline cellulose oral
Drug: XPF-010 — Capsule filled with XEN1101
  Arms: Drug: XEN1101 XPF-008 Formulation Oral Drug: XEN1101 XPF-010 Formulation Oral; Drug: XEN1101 XPF-010 Formulation Oral
Drug: Itraconazole 400mg — Oral
  Arms: Drug: XEN1101 XPF-010 Formulation Oral Drug: Itraconazole 400mg Oral

SUMMARY:
The XEN1101 Phase 1 clinical trial is a randomized, double-blind, placebo-controlled study that will evaluate the safety, tolerability and PK of both single ascending doses (SAD) and multiple ascending doses (MAD) of XEN1101 in healthy subjects. In addition to safety and PK data, the clinical trial has been designed to include a pharmacodynamic read-out by incorporating a pilot transcranial magnetic stimulation (TMS) sub-study. The TMS model sub-study is designed to demonstrate delivery of XEN1101 into the central nervous system and to observe a change in cortical excitability as measured by EEG and/or electromyographic (EMG) activity.

Part 3, 4 and 5: Phase 1, randomised, multi part study to evaluate the safety, tolerability, PK, relative bioavailability and food effect of single and multiple ascending doses of XEN1101 and Preliminary Drug-Drug Interaction Assessment with Itraconazole.

DETAILED DESCRIPTION:
Part 1 will study safety, tolerability, PK of single ascending doses (SAD) of XPF-008 as well as the impact and variability of single ascending doses of XPF-008 on TMS.

Part 2 will study the safety, tolerability and PK of multiple ascending doses (MAD) of XPF-008

Part 3 will explore dose proportionality of XPF-010 and confirm dosing for subsequent cohorts, and the food effect and relative bioavailability of XPF-010 compared to XPF-008.

Part 4 will explore multiple dose PK.

Part 5 will explore the drug-drug interaction of XPF-010, when given with itraconazole.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or females aged between 18 and 55 years inclusive with a body mass index (BMI) between 18.50 and 30.00 kg/m2
* Must agree to use effective methods of contraception, if applicable
* Able to swallow capsules
* Able to provide written, personally signed and dated informed consent form (ICF)

Key Exclusion Criteria:

* Any history of epileptic seizures
* Any current and relevant history of significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk, affect clinical or laboratory results, or the subject's ability to participate in the study
* Answering "yes" to any of the questions within the Columbia Suicide Severity Rating Scale
* Mental incapacity or lingual barriers precluding adequate understanding, cooperation, and compliance with the study
* No prescription or over-the-counter (OTC) medications (except hormonal contraception), herbal or dietary supplements OTC medications 14 days prior to dosing to study end
* No smoking 60 days prior to dosing to study end
* No soft drugs 3 months prior to Screening and hard drugs 2 years prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Parts 1 & 2: Number of Participants with Adverse Events (AEs) | From screening (28 days prior to Day 1) through to 30 days post-final dose
  To assess AEs as a criteria of safety and tolerability
Parts 1 & 2: Resting electrocardiogram (ECG) | At screening (28 days prior to Day 1) through to 7 days post-final dose
  To assess ECG as a criteria of safety and tolerability
Parts 1 & 2: Vital signs | At screening (28 days prior to Day 1) through to 7 days post-final dose
  To assess vital signs as a criteria of safety and tolerability
Part 3a: Maximum Observed Plasma Concentration (Cmax) of XEN1101 | At screening (27 days prior to Day -1) through to 31 days post dose
  To characterize the PK profile of XEN1101 and M11 (a metabolite of XEN1101) in plasma of single ascending, oral doses of XPF-010
Part 3a: Area under the plasma concentration-time curve (AUC) of XEN1101 | At screening (27 days prior to Day -1) through to 31 days post dose
  To characterize the PK profile of XEN1101 and M11 (a metabolite of XEN1101) in plasma of single ascending, oral doses of XPF-010
Part 3a: Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations | At screening (27 days prior to Day -1) through to 31 days post dose
  To evaluate the safety and tolerability of XEN1101 (XPF-010)
Part 3b: Maximum Observed Plasma Concentration (Cmax) of XEN1101 | At screening (27 days prior to Day -1) through to 31 days post dose
  To assess the Food Effect on PK (Cmax) and the relative bioavailability/comparability (Cmax) of XEN1101 following single oral doses of XPF-010 (fed), XPF-008 (fed) and XPF-010 (fasted)
Part 3b: Area under the plasma concentration-time curve (AUC) of XEN1101 | At screening (27 days prior to Day -1) through to 31 days post dose
  To assess the Food Effect on PK (AUC0-240h) and the relative bioavailability/comparability (AUC0-240h) of XEN1101 following single oral doses of XPF-010 (fed), XPF-008 (fed) and XPF-010 (fasted)
Part 3b: Frequency and severity of TEAEs, treatment-emergent SAEs, and TEAEs leading to treatment discontinuations | At screening (27 days prior to Day -1) through to 31 days post dose
  To evaluate the safety and tolerability of XEN1101
Part 4: Maximum Observed Plasma Concentration (Cmax) of XEN1101 | At screening (27 days prior to Day -1) through to 51 days post dose
  To characterize the PK profile of XEN1101 and M11 (metabolite of XEN1101) in plasma of multiple daily oral doses of XPF-010
Part 4: Area under the plasma concentration-time curve (AUC) of XEN1101 | At screening (27 days prior to Day -1) through to 51 days post dose
  To characterize the PK profile of XEN1101 and M11 (metabolite of XEN1101) in plasma of multiple daily oral doses of XPF-010
Part 4: Frequency and severity of TEAEs, treatment-emergent SAEs, and TEAEs leading to treatment discontinuations | At screening (27 days prior to Day -1) through to 51 days post dose
  To evaluate the safety and tolerability of XEN1101 (XPF-010)
Part 5: Maximum Observed Plasma Concentration (Cmax) of XEN1101 | Day 10 and Day 11
  To assess the PK of XEN1101 (XPF-010) in the presence and absence of itraconazole
Part 5: Area under the plasma concentration-time curve (AUC) of XEN1101 | Day 10 and Day 11
  To assess the PK of XEN1101 (XPF-010) in the presence and absence of itraconazole
Part 5: Frequency and severity of TEAEs, treatment-emergent SAEs, and TEAEs leading to treatment discontinuations | At screening (27 days prior to Day -1) through to 51 days post dose
  To evaluate the safety and tolerability of XEN1101 (XPF-010)

SECONDARY OUTCOMES:
Parts 1 & 2: Maximum Observed Plasma Concentration (Cmax) | Day 1 predose through to 7 days post-final dose
  Cmax is the maximum observed plasma concentration in ng/mL
Parts 1 & 2: Time to the Maximum Observed Plasma Concentration (Tmax) | Day 1 predose through to 7 days post-final dose
  Tmax is the time in hours to reach Cmax following dosing
Parts 1 & 2: Terminal elimination half-life (t1/2) | Day 1 predose through to 7 days post-final dose
  The time in hours required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase
Parts 1 & 2: Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Quantifiable Plasma Concentration (AUC0-last) | Day 1 predose through to 7 days post-final dose
  The area under the plasma concentration-time curve [in ng.h/mL] from time zero to the time corresponding to the last quantifiable plasma concentration
Parts 3 to 5: Cardiac Safety | At screening (27 days prior to Day -1) through to 11 days post dose for Parts 3a and 3b and at screening (27days prior to Day -1) through to Day 21
  To evaluate the cardiovascular safety profile of XEN1101 (XPF-010), assessing potential ECG interval changes from baseline following dosing, in particular any effects on the QTc interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory N Beatch, PhD, Study Director — Xenon Pharmaceuticals Inc.
Locations (1):
- Richmond Pharmacology Ltd., London, United Kingdom